CLINICAL TRIAL: NCT05792709
Title: Effects of Oral Motor Therapy in Children With Cerebral Palsy ; A Randomized Control Trial
Brief Title: Effects of Oral Motor Therapy in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Principal Investigator, Hafiza Shabnum Noor, Senior Lecturer, Riphah International University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0646
Record Dates: First submitted 2023-02-26; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Cerebral Palsy
Keywords: Oral Motor Therapy; Cerebral palsy; Drooling scale; Feeding and Swallowing
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Masking Description: All patients of study were screened for following information before randomization such as age, gender, location duration of disease and medical history. Each participant of current study was undergoing through questionnaire regarding demographic information. For oral motor therapy assessment and the Functional Feeding Assessment (FFA) subscale of the multidisciplinary Feeding Profile (MFP) were used. A blinded pedagogue who was not involve in the training sessions performed the Bayley scales of infant development (BSID-II) before and after the training.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Motor Therapy (Experimental): These are exercises designed to increase the range of movement in tongue, lips, and jaw, which helped in speech and/or swallow functioning. It is important to move the designated area as far as can in each direction until feel the muscles stretch. Stop if feel any pain, and mention it to speech therapist or doctor. Practice these exercises, once through, 10 times a day.
  Interventions: Other: Oral Motor Therapy
- Traditional Therapy (Other): weeks traditional Speech Therapy was provided. Pre-language skills (vocalizations) manual sign languages, gestures, picture communication boards, voice output communication devices were used. Playing and talking, using pictures, books, objects, or ongoing events to help language development. Use of repetition exercises to build speech and language skills.
  Interventions: Other: Oral Motor Therapy

INTERVENTIONS:
Other: Oral Motor Therapy — In Traditional therapy we will give cognitive and articulation therapy to the patients.
  Other Names: Traditional Therapy

SUMMARY:
: CP is a neurodevelopmental condition. A set of irreversible impairments of movement and posture development, resulting in activity limitation. Acquired CP can be the outcome of a variety of issues that arise after the first 28 days of a baby's existence. A CP diagnosis can now be made as early as 16 weeks. speech-language pathologists (SLPs) began collaborating with OTs and PTs for Infants and toddlers who also struggle with speech impediments, feeding and swallowing disorder. Oral motor exercises (OMEs), also known as "mouth exercises," "non-speech oral motor training," and "oral motor treatment" were designed for their treatment. The objective of this study was to assess the effects of oral motor exercises in children with cerebral palsy having feeding and swallowing difficulties.

DETAILED DESCRIPTION:
Over 17 million people throughout the world are living with cerebral palsy (CP), making it the most common physical disability among children. CP is a neurodevelopmental condition[1]. Cerebral palsy is a fitting classification of the condition and its associated deficits because the word cerebral means "pertaining to the brain" and palsy means "loss of muscle control." A set of irreversible impairments of movement and posture development, resulting in activity limitation, that are linked to non-progressive disruptions that occurred in the developing foetus or infant brain, was chosen as the official definition of CP in 2005 by the International Consensus [2]. It's important to keep in mind that the phrase "cerebral palsy" refers to a spectrum of conditions, each of which has its own unique appearance, set of symptoms, and prevalence rate within the general population. In addition to the musculoskeletal and neurological symptoms of CP, epilepsy and other sensory and cognitive impairments are also common

ELIGIBILITY:
Inclusion Criteria:

1. CP children already diagnosed with feeding and swallowing difficulties.
2. Age range: 4 to13 years

Exclusion Criteria:

1. Patients with any co morbid conditions like uncontrolled epilepsy.
2. Patients on NG or feeding tube.

Ages: 4 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2022-08-16 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-02-27 (Actual)

PRIMARY OUTCOMES:
Feeding Oral Motor scale | upto 16 weeks
  This tool is used to evaluate the posture, jaw mobility, tongue activity, lips, feeding behavior, abnormal reflexes and breathing control

SECONDARY OUTCOMES:
Drooling severity and frequency scale | upto 24 weeks
  This tool is used to check the severity of drooling

CONTACTS AND LOCATIONS:
Overall Officials: Ghazal Awais, MS-SLP, Principal Investigator — Riphah International University; Hafiza Shabnum Noor, MS-SLP, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Hafiza Shabnum Noor, Lahore, Punjab Province
  - Hafiza Shabnum Noor, Lahore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Turra GS, Schwartz IVD, Almeida ST, Martinez CC, Bridi M, Barreto SSM. Efficacy of speech therapy in post-intubation patients with oropharyngeal dysphagia: a randomized controlled trial. Codas. 2021 Apr 26;33(2):e20190246. doi: 10.1590/2317-1782/20202019246. eCollection 2021. PMID 33909759
- [Background] Sigan SN, Uzunhan TA, Aydinli N, Eraslan E, Ekici B, Caliskan M. Effects of oral motor therapy in children with cerebral palsy. Ann Indian Acad Neurol. 2013 Jul;16(3):342-6. doi: 10.4103/0972-2327.116923. PMID 24101813
- See also: Study Protocol — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3788277/
- Available data/document: Study Protocol — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3788277/